CLINICAL TRIAL: NCT00500266
Title: A Phase 3, Open-Label, Single-Arm Trial Evaluating the Safety, Tolerability, & Reactogenicity of a 13vPnC Vaccine in Ambulatory Elderly Adults Aged 68 Years & Older Who Received 1 or More Doses of 23vPS Vaccine at Least 3 Years Before Study Enrollment
Brief Title: Study Evaluating Safety of 13-Valent Pneumococcal Conjugate Vaccine in Healthy Elderly Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 6115A1-3000
Record Dates: First submitted 2007-07-09; First posted 2007-07-11 (Estimated); Results first posted 2011-09-16 (Estimated); Last update posted 2011-09-16 (Estimated); Status verified 2011-08

CONDITIONS: Pneumococcal Infections
Keywords: pneumococcal conjugate vaccine; vaccine
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): 13-valent Pneumococcal Conjugate Vaccine
  Interventions: Biological: 13-valent Pneumococcal Conjugate Vaccine (13vPnC)

INTERVENTIONS:
Biological: 13-valent Pneumococcal Conjugate Vaccine (13vPnC)

SUMMARY:
To evaluate the safety of 13-valent pneumococcal conjugate vaccine (13vPnC) in elderly subjects who were vaccinated with one or more doses of 23-valent pneumococcal polysaccharide vaccine (23vPS) at least 3 years before study enrollment.

ELIGIBILITY:
MAIN INCLUSION CRITERIA:

* Male or female aged 68 years or older
* Determined by medical history, physical examination, and clinical judgment to be eligible for the study
* Documented vaccination with 1 or more doses of pneumococcal vaccine at least 3 years before study enrollment

MAIN EXCLUSION CRITERIA:

* Known history of severe reaction to a vaccine
* Documented S pneumoniae infection within the past 5 years.
* Known or suspected immunodeficiency or receiving treatment with immunosuppressive therapy including cytotoxic agents or systemic corticosteroids
* Serious chronic disorder including metastatic malignancy, severe chronic obstructive pulmonary disease requiring supplemental oxygen, end-stage renal disease with or without dialysis, clinically unstable cardiac disease, or any other disorder that in the investigator's opinion precludes the subject from participating in the study.

Min Age: 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1053 (Actual)
Dates: Start 2008-05; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (54):
- United States (36):
  - Chandler, Arizona
  - Glendale, Arizona
  - Phoenix, Arizona
  - Rolling Hills Estates, California
  - Apopka, Florida
  - Boynton Beach, Florida
  - Chiefland, Florida
  - Gainesville, Florida
  - Largo, Florida
  - Melbourne, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Arkansas City, Kansas
  - Newton, Kansas
  - Wichita, Kansas
  - Crescent Springs, Kentucky
  - New Orleans, Louisiana
  - Nitchitoches, Louisiana
  - Camillus, New York
  - Rochester, New York
  - Raleigh, North Carolina
  - Akron, Ohio
  - Canal Fulton, Ohio
  - Columbus, Ohio
  - Franklin, Ohio
  - Portland, Oregon
  - Pittsburgh, Pennsylvania
  - Goose Creek, South Carolina
  - Mt. Pleasant, South Carolina
  - Houston, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - West Jordan, Utah
  - Bellingham, Virginia
  - Walla Walla, Washington
  - Wenatchee, Washington
- Germany (11):
  - Berlin
  - Berlin-Wilmersdorf
  - Charlottenburg
  - Deggingen
  - Frankfurt am Main
  - Hanover
  - Kassel
  - Leipzig
  - Offenbach
  - Wangen
  - Würzburg
- Sweden (7):
  - Arlöv
  - Gothenburg
  - Skene
  - Skivarp
  - Stockholm
  - Umeå
  - Uppsala

RESULTS

PARTICIPANT FLOW:
Groups:
- 13vPnC: Participants received single 0.5 milliliter (mL) dose of 13-valent pneumococcal conjugate vaccine (13vPnC) into the deltoid muscle of the arm.
Period: Overall Study
Arm/Group | 13vPnC
Started | 1053
Treated | 1049
Completed | 1040
Not Completed | 13
Not completed — Death | 3
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 3
Not completed — Assigned, not treated | 4

BASELINE CHARACTERISTICS:
Arm/Group | 13vPnC
Number analyzed (Participants) | 1049
Age Continuous [Mean (Standard Deviation); unit: years] | 75.3 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 584
  Male | 465

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Pre-specified Local Reactions
Description: Local reactions were collected by the participant using an electronic diary. Redness and swelling scaled as any(present); mild(2.5-5.0 centimeters[cm]); moderate(5.1-10.0 cm); severe(>10.0cm). Pain as any(present); mild(present, no interference with activity); moderate(present, some interference with activity); severe(present, prevents daily activity). Limitation of arm movement as any(present); mild(present, could move arm above head); moderate(could move arm above shoulder but not above head); severe(could not move arm above shoulder). Participants may be represented in more than 1 category.
Time Frame: Days 1 through 14
Population: Safety population: all participants who received 1 dose of 13vPnC. n = participants reporting "yes" for at least 1 day or "no" for all days.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 13vPnC
Number analyzed (Participants) | 1049
Percentage of Participants
  Redness: Any (n=666) | 14.3 [11.7 to 17.2]
  Redness: Mild (n=660) | 12.6 [10.1 to 15.3]
  Redness: Moderate (n=649) | 6.5 [4.7 to 8.6]
  Redness: Severe (n=638) | 1.1 [0.4 to 2.2]
  Swelling: Any (n=664) | 12.8 [10.4 to 15.6]
  Swelling: Mild (n=658) | 10.9 [8.7 to 13.6]
  Swelling: Moderate (n=651) | 5.5 [3.9 to 7.6]
  Swelling: Severe (n=636) | 0.6 [0.2 to 1.6]
  Pain: Any (n=777) | 51.0 [47.4 to 54.5]
  Pain: Mild (n=770) | 49.4 [45.8 to 52.9]
  Pain: Moderate (n=656) | 9.0 [6.9 to 11.4]
  Pain: Severe (n=634) | 0.2 [0.0 to 0.9]
  Limitation of arm movement: Any (n=679) | 16.2 [13.5 to 19.2]
  Limitation of arm movement: Mild (n=674) | 14.8 [12.2 to 17.7]
  Limitation of arm movement: Moderate (n=636) | 1.6 [0.8 to 2.9]
  Limitation of arm movement: Severe (n=640) | 1.6 [0.8 to 2.9]
  Any local reaction (n=802) | 56.6 [53.1 to 60.1]
  Any severe local reaction (n=643) | 2.6 [1.5 to 4.2]

2. Primary Outcome: Percentage of Participants With Pre-specified Systemic Events
Description: Systemic events were collected by participant using electronic diary. Fatigue,headache,new/aggravated generalized muscle pain,new/aggravated generalized joint pain: any, mild(no interference with activity), moderate(some interference with activity), severe(prevents routine daily activity). Fever(>=38 degrees Celsius[C]), chills, rash, vomiting(mild:1-2 times daily; moderate:>2 times daily; severe:prevents daily activity) decreased appetite & diarrhea(mild:2-3 loose stools/day; moderate:4-5 loose stools/day; severe:>=6 loose stools/day) reported. Participants may be represented in >1 category.
Time Frame: Days 1 through 14
Population: Safety population: all participants who received 1 dose of 13vPnC. n = number of participants with the event as "yes" for at least 1 day or as "no" for all days.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 13vPnC
Number analyzed (Participants) | 1049
Percentage of Participants
  Fever (any): >=38 degrees C (n=641) | 2.0 [1.1 to 3.4]
  Fever: >=38 degrees C but <38.5 degrees C (n=636) | 0.8 [0.3 to 1.8]
  Fever: >=38.5 degrees C but <39 degrees C (n=634) | 0.0 [0.0 to 0.6]
  Fever: >=39 degrees C but <=40 degrees C (n=635) | 0.3 [0.0 to 1.1]
  Fever: >40 degrees C (n=638) | 0.9 [0.3 to 2.0]
  Fatigue: Any (n=733) | 34.4 [30.9 to 37.9]
  Fatigue: Mild (n=710) | 28.7 [25.4 to 32.2]
  Fatigue: Moderate (n=683) | 15.2 [12.6 to 18.1]
  Fatigue: Severe (n=639) | 2.0 [1.1 to 3.5]
  Headache: Any (n=702) | 26.1 [22.9 to 29.5]
  Headache: Mild (n=696) | 24.1 [21.0 to 27.5]
  Headache: Moderate (n=655) | 9.0 [6.9 to 11.5]
  Headache: Severe (n=637) | 0.8 [0.3 to 1.8]
  Chills (n=651) | 7.5 [5.6 to 9.8]
  Rash (n=658) | 8.4 [6.4 to 10.7]
  Vomiting: Any (vomiting present; n=638) | 0.9 [0.3 to 2.0]
  Vomiting: Mild (1 to 2 times in 24 hours;n=637) | 0.8 [0.3 to 1.8]
  Vomiting: Moderate (>2 times in 24 hours;n=635) | 0.2 [0.0 to 0.9]
  Vomiting: Severe (prevents routine activity;n=634) | 0.0 [0.0 to 0.6]
  Decreased appetite (n=668) | 11.2 [8.9 to 13.9]
  Diarrhea: Any (diarrhea present; n=684) | 14.5 [11.9 to 17.3]
  Diarrhea: Mild (2 to 3 loose stools/day; n=678) | 12.8 [10.4 to 15.6]
  Diarrhea: Moderate (4 to 5 loose stools/day;n=644) | 3.4 [2.2 to 5.1]
  Diarrhea: Severe (>=6 loose stools/day; n=635) | 0.3 [0.0 to 1.1]
  New generalized muscle pain: Any (n=700) | 25.3 [22.1 to 28.7]
  New generalized muscle pain: Mild (n=679) | 20.5 [17.5 to 23.7]
  New generalized muscle pain: Moderate (n=658) | 7.9 [6.0 to 10.2]
  New generalized muscle pain: Severe (n=636) | 0.6 [0.2 to 1.6]
  Aggravated generalized muscle pain: Any (n=669) | 12.3 [9.9 to 15.0]
  Aggravated generalized muscle pain: Mild (n=650) | 7.5 [5.6 to 9.8]
  Aggravated generalized muscle pain:Moderate(n=655) | 6.4 [4.7 to 8.6]
  Aggravated generalized muscle pain: Severe (n=639) | 1.4 [0.6 to 2.7]
  New generalized joint pain: Any (n=665) | 12.8 [10.3 to 15.6]
  New generalized joint pain: Mild (n=651) | 8.1 [6.2 to 10.5]
  New generalized joint pain: Moderate (n=648) | 5.7 [4.1 to 7.8]
  New generalized joint pain: Severe (n=637) | 0.8 [0.3 to 1.8]
  Aggravated generalized joint pain: Any (n=661) | 9.7 [7.5 to 12.2]
  Aggravated generalized joint pain: Mild (n=647) | 5.7 [4.1 to 7.8]
  Aggravated generalized joint pain: Moderate(n=647) | 5.1 [3.5 to 7.1]
  Aggravated generalized joint pain: Severe (n=637) | 1.1 [0.4 to 2.3]
  Any systemic event (n=832) | 58.4 [55.0 to 61.8]

3. Primary Outcome: Percentage of Participants Taking Pain or Antipyretic Medication
Description: Use of pain or antipyretic medication was collected by the participants using an electronic diary.
Time Frame: Days 1 through 14
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 13vPnC
Number analyzed (Participants) | 1049
Percentage of Participants
  Use of medication to treat pain (n=677) | 17.0 [14.2 to 20.0]
  Use of medication to treat fever (n=655) | 6.4 [4.7 to 8.6]

ADVERSE EVENTS:
Time Frame: Local reactions, systemic events recorded within 14 days post vaccination. AEs recorded from Visit(V) 1 to 2(29-43 days after V1). At V3(166-194 days after V1), only newly diagnosed chronic medical conditions recorded as AEs. SAEs recorded from V1 to V3.
Description: Local reactions and systemic events were collected by the participants using an electronic diary checklist (systematic assessment). AE/SAEs were documented by investigator on the case report form (non-systematic assessment) at each visit.
Groups:
- 13vPnC: Visit 1 to Visit 2: Participants received a single 0.5 mL dose of 13vPnC into the deltoid muscle of the arm once during the study. Local reactions and systemic events were collected from Day 1 through Day 14. AEs were recorded from Visit 1 to Visit 2 (29-43 days after Visit 1). SAEs were collected throughout the study.
- 13vPnC: 6-month Follow-up: Participants received a single 0.5 mL dose of 13vPnC into the deltoid muscle of the arm once during the study. At visit 3, the 6-month follow-up (166-194 days after Visit 1) only newly diagnosed chronic medical conditions were collected as AEs. SAEs were collected throughout the study.
Arm/Group | 13vPnC: Visit 1 to Visit 2 | 13vPnC: 6-month Follow-up
Serious Adverse Events (participants affected / at risk) | 10/1049 | 41/1049
Other Adverse Events (participants affected / at risk) | 486/1049 | 77/1049
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 13vPnC: Visit 1 to Visit 2 (N=1049) | 13vPnC: 6-month Follow-up (N=1049)
Bradyarrhythmia (Cardiac disorders) | 1 | 1
Tachyarrhythmia (Cardiac disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 3
Atrial fibrillation (Cardiac disorders) | 0 | 2
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 3
Abscess limb (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Enteritis infectious (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Fracture displacement (Injury, poisoning and procedural complications) | 0 | 1
Postoperative renal failure (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Fibrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Guillain-Barre syndrome (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Percutaneous coronary intervention (Surgical and medical procedures) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 13vPnC: Visit 1 to Visit 2 (N=1049) | 13vPnC: 6-month Follow-up (N=1049)
Redness (any) (Skin and subcutaneous tissue disorders) | 95/666 | 0/0 — Redness (any) = present at site of vaccination.
Redness (mild) (Skin and subcutaneous tissue disorders) | 83/660 | 0/0 — Redness (mild) = 2.5 to 5.0 cm
Redness (moderate) (Skin and subcutaneous tissue disorders) | 42/649 | 0/0 — Redness (moderate) = 5.1 to 10.0 cm
Redness (severe) (Skin and subcutaneous tissue disorders) | 7/638 | 0/0 — Redness (severe) = >10.0 cm
Swelling (any) (Skin and subcutaneous tissue disorders) | 85/664 | 0/0 — Swelling (any) = present at site of vaccination
Swelling (mild) (Skin and subcutaneous tissue disorders) | 72/658 | 0/0 — Swelling (mild) = 2.5 to 5.0 cm
Swelling (moderate) (Skin and subcutaneous tissue disorders) | 36/651 | 0/0 — Swelling (moderate) = 5.1 to 10.0 cm
Swelling (severe) (Skin and subcutaneous tissue disorders) | 4/636 | 0/0 — Swelling (severe) = 10.0 cm
Pain (any) (Skin and subcutaneous tissue disorders) | 396/777 | 0/0 — Pain (any) = present at site of vaccination.
Pain (mild) (Skin and subcutaneous tissue disorders) | 380/770 | 0/0 — Pain (mild) = no interference with activity.
Pain (moderate) (Skin and subcutaneous tissue disorders) | 59/656 | 0/0 — Pain (moderate) = some interference with activity.
Pain (severe) (Skin and subcutaneous tissue disorders) | 1/634 | 0/0 — Pain (severe) = prevents routine daily activity.
Limitation of arm movement (any) (Skin and subcutaneous tissue disorders) | 110/679 | 0/0 — Limitation of arm movement (any) = present due to vaccination.
Limitation of arm movement (mild) (Skin and subcutaneous tissue disorders) | 100/674 | 0/0 — Limitation of arm movement (mild) = some limitation of arm movement.
Limitation of arm movement (moderate) (Skin and subcutaneous tissue disorders) | 10/636 | 0/0 — Limitation of arm movement (moderate) = unable to move arm above head but able to move arm above shoulder.
Limitation of arm movement (severe) (Skin and subcutaneous tissue disorders) | 10/640 | 0/0 — Limitation of arm movement (severe) = unable to move arm above shoulder.
Fever (any) (General disorders) | 13/641 | 0/0 — Fever (any) = ≥38 degrees C
Fever (mild) (General disorders) | 5/636 | 0/0 — Fever (mild) = ≥38 degrees C but <38.5 degrees C
Fever (moderate) (General disorders) | 0/634 | 0/0 — Fever (moderate) = ≥38.5 degrees C but <39 degrees C.
Fever (severe) (General disorders) | 2/635 | 0/0 — Fever (severe) = ≥39 degrees C but ≤40 degrees C
Fever (potentially life threatening) (General disorders) | 6/638 | 0/0 — Fever (potentially life threatening) = >40 degrees C
Fatigue (any) (General disorders) | 252/733 | 0/0 — Fatigue (any) = fatigue present
Fatigue (mild) (General disorders) | 204/710 | 0/0 — Fatigue (mild) = no interference with activity.
Fatigue (moderate) (General disorders) | 104/683 | 0/0 — Fatigue (moderate) = some interference with activity.
Fatigue (severe) (General disorders) | 13/639 | 0/0 — Fatigue (severe) = prevents routine daily activity.
Headache (any) (General disorders) | 183/702 | 0/0 — Headache (any) = headache present.
Headache (mild) (General disorders) | 168/696 | 0/0 — Headache (mild) = no interference with activity.
Headache (moderate) (General disorders) | 59/655 | 0/0 — Headache (moderate) = some interference with activity.
Headache (severe) (General disorders) | 5/637 | 0/0 — Headache (severe) = prevents routine daily activity.
Chills (General disorders) | 49/651 | 0/0
Rash (General disorders) | 55/658 | 0/0
Vomiting (any) (General disorders) | 6/638 | 0/0 — Vomiting (any) = vomiting present.
Vomiting (mild) (General disorders) | 5/637 | 0/0 — Vomiting (mild) = no interference with activity or 1 to 2 times in 24 hours.
Vomiting (moderate) (General disorders) | 1/635 | 0/0 — Vomiting (moderate) = some interference with activity or more than 2 times in 24 hours.
Vomiting (severe) (General disorders) | 0/634 | 0/0 — Vomiting (severe) = prevents routine daily activity.
Decreased appetite (General disorders) | 75/668 | 0/0
Diarrhea (any) (General disorders) | 99/684 | 0/0 — Diarrhea (any) = diarrhea present.
Diarrhea (mild) (General disorders) | 87/678 | 0/0 — Diarrhea (mild) = 2 to 3 loose stools in 24 hours.
Diarrhea (moderate) (General disorders) | 22/644 | 0/0 — Diarrhea (moderate) = 4 to 5 loose stools in 24 hours.
Diarrhea (severe) (General disorders) | 2/635 | 0/0 — Diarrhea (severe) = 6 or more loose stools in 24 hours.
New generalized muscle pain (any) (General disorders) | 177/700 | 0/0 — New generalized muscle pain (any) = new generalized muscle pain present.
New generalized muscle pain (mild) (General disorders) | 139/679 | 0/0 — New generalized muscle pain (mild) = no interference with activity.
New generalized muscle pain (moderate) (General disorders) | 52/658 | 0/0 — New generalized muscle pain (moderate) = some interference with activity.
New generalized muscle pain (severe) (General disorders) | 4/636 | 0/0 — New generalized muscle pain (severe) = prevents routine daily activity.
Aggravated generalized muscle pain (any) (General disorders) | 82/669 | 0/0 — Aggravated generalized muscle pain (any) = aggravated generalized muscle pain present.
Aggravated generalized muscle pain (mild) (General disorders) | 49/650 | 0/0 — Aggravated generalized muscle pain (mild) = no interference with activity.
Aggravated generalized muscle pain (moderate) (General disorders) | 42/655 | 0/0 — Aggravated generalized muscle pain (moderate) = some interference with activity.
Aggravated generalized muscle pain (severe) (General disorders) | 9/639 | 0/0 — Aggravated generalized muscle pain (severe) = prevents routine daily activity.
New generalized joint pain (any) (General disorders) | 85/665 | 0/0 — New generalized joint pain (any) = new generalized joint pain present.
New generalized joint pain (mild) (General disorders) | 53/651 | 0/0 — New generalized joint pain (mild) = no interference with activity.
New generalized joint pain (moderate) (General disorders) | 37/648 | 0/0 — New generalized joint pain (moderate) = some interference with activity.
New generalized joint pain (severe) (General disorders) | 5/637 | 0/0 — New generalized joint pain (severe) = prevents routine daily activity.
Aggravated generalized joint pain (any) (General disorders) | 64/661 | 0/0 — Aggravated generalized joint pain (any) = aggravated generalized joint pain present.
Aggravated generalized joint pain (mild) (General disorders) | 37/647 | 0/0 — Aggravated generalized joint pain (mild) = no interference with activity.
Aggravated generalized joint pain (moderate) (General disorders) | 33/647 | 0/0 — Aggravated generalized joint pain (moderate) = some interference with activity.
Aggravated generalized joint pain (severe) (General disorders) | 7/637 | 0/0 — Aggravated generalized joint pain (severe) = prevents routine daily activity.
Bradycardia (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Blepharitis (Eye disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 0
Diabetic retinopathy (Eye disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 6 | 0
Nausea (Gastrointestinal disorders) | 6 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0
Constipation (Gastrointestinal disorders) | 2 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0
Retching (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 4 | 1
Injection site pain (General disorders) | 2 | 0
Injection site haematoma (General disorders) | 1 | 0
Injection site pruritus (General disorders) | 1 | 0
Injection site swelling (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Pain (General disorders) | 1 | 1
Seasonal allergy (Immune system disorders) | 1 | 0
Bronchitis (Infections and infestations) | 6 | 1
Sinusitis (Infections and infestations) | 4 | 1
Upper respiratory tract infection (Infections and infestations) | 4 | 0
Urinary tract infection (Infections and infestations) | 4 | 1
Gastroenteritis (Infections and infestations) | 2 | 0
Gastroenteritis viral (Infections and infestations) | 2 | 0
Herpes zoster (Infections and infestations) | 2 | 0
Acute sinusitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Ear infection (Infections and infestations) | 1 | 0
Eye infection (Infections and infestations) | 1 | 0
Laryngitis (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 1 | 0
Nail infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Staphylococcal skin infection (Infections and infestations) | 1 | 0
Tinea cruris (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 1
Skin laceration (Injury, poisoning and procedural complications) | 3 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 1
Limb injury (Injury, poisoning and procedural complications) | 2 | 0
Electric shock (Injury, poisoning and procedural complications) | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Joint sprain (Injury, poisoning and procedural complications) | 1 | 0
Blood glucose increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 5
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 3
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 1
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endobronchial lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dizziness (Nervous system disorders) | 3 | 0
Headache (Nervous system disorders) | 3 | 0
Paraesthesia (Nervous system disorders) | 3 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0
Polyneuropathy (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Bipolar disorder (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 2
Stress (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Bladder spasm (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 1
Skin mass (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 3 | 3
Hypotension (Vascular disorders) | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 1
Aortic valve incompetence (Cardiac disorders) | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Left ventricular hypertrophy (Cardiac disorders) | 0 | 1
Tricuspid valve incompetence (Cardiac disorders) | 0 | 1
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 3
Diverticulum (Gastrointestinal disorders) | 0 | 2
Haemorrhoids (Gastrointestinal disorders) | 0 | 2
Pain (General disorders) | 0 | 1
Suprapubic pain (General disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Oral herpes (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Blood thyroid stimulating hormone increased (Investigations) | 0 | 1
Cardiac murmur (Investigations) | 0 | 1
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 3
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 2
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Narcolepsy (Nervous system disorders) | 0 | 1
Restless legs syndrome (Nervous system disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Hypertonic bladder (Renal and urinary disorders) | 0 | 1
Renal mass (Renal and urinary disorders) | 0 | 1
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Milia (Skin and subcutaneous tissue disorders) | 0 | 1
Joint prosthesis user (Social circumstances) | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 0 | 1
Temporal arteritis (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.